CLINICAL TRIAL: NCT00163592
Title: Non- Interventional Study of Tissucol® for Hemostasis in Subjects With Femoral Vascular Anastomosis Undergoing Vascular Reconstruction With PTFE Prosthesis
Brief Title: Post-Marketing Surveillance of TISSUCOL for Hemostasis in Subjects Undergoing Vascular Reconstruction With Polytetrafluoroethylene (PTFE) Prosthesis
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Other Study IDs: 530301
Record Dates: First submitted 2005-09-08; First posted 2005-09-14 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Femoral Vascular Anastomosis
Keywords: Vascular reconstruction; Polytetraflouroethylene (PTFE) prosthesis
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Drug: Tissucol®
Procedure: Control: Conventional treatment, i.e. compression with swabs

SUMMARY:
This study investigates if the time to hemostasis can be reduced by application of Tissucol® onto femoral vascular anastomoses with PTFE prostheses compared to standard methods, such as compression with swabs.

ELIGIBILITY:
Subjects with femoral vascular anastomosis and bleeding suture holes after vessel reconstruction with a PTFE prosthesis

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bürger, MD, Principal Investigator — University Clinics of Magdeburg, Germany
Locations (5):
- Austria (2):
  - General Hospital (AKH) Salzburg, Salzburg, Salzburg
  - Landeskrankenhaus Innsbruck, Innsbruck, Tyrol
- Germany (3):
  - Leonberg Hospital, Department of Vascular Surgery, Leonberg
  - University Clinics of Magdeburg, Department of Vascular Surgery, Magdeburg
  - Klinikum Nürnberg Süd, Department of Vascular Surgery, Nuremberg